CLINICAL TRIAL: NCT04183166
Title: A Randomized Phase I/II Trial in Patients With Newly Diagnosed, Locoregionally Advanced Squamous Cell Carcinoma of the Head and Neck (SCCHN) Evaluating a Mutanome-directed Immunotherapy.
Brief Title: A Clinical Trial Evaluating TG4050 in Head and Neck Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Transgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TG4050.02
Record Dates: First submitted 2019-11-21; First posted 2019-12-03 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A : Early study treatment initiation (Experimental): TG4050 treatment initiation at completion of primary treatment
  Interventions: Drug: TG4050
- Arm B: Study treatment initiation at recurrence (Experimental): TG4050 treatment initiation at the time of recurrence
  Interventions: Drug: TG4050

INTERVENTIONS:
Drug: TG4050 — Subcutaneous injections weekly for the first 6 weeks and then every 3 weeks

SUMMARY:
This is a multicenter, open-label, two arms, randomized, phase I/II study evaluating the safety and tolerability as well as some activity parameters of TG4050 in patients with squamous cell carcinoma of the head and neck (SCCHN).

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Newly diagnosed stage III or IV, amenable to surgery (AJCC 8th edition) squamous-cell carcinoma of the oral cavity, oropharynx, hypopharynx or larynx
3. Female or male patients, aged at least 18 years
4. Patients in Complete Response after treatment of their primary tumor.
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.
6. Adequate hematological, hepatic and renal functions

Exclusion Criteria:

1. Patients with carcinoma of the nasopharynx, squamous cell-carcinoma of unknown primary, squamous cell carcinoma that originates from the skin and salivary gland or paranasal sinus, non-squamous histologies.
2. Prior exposure to anti-cancer vaccines and any antibody targeting T-cell co-regulatory proteins such as anti-PD1, anti-PDL1 or anti-CTLA4 antibodies.
3. Other active malignancy requiring concurrent systemic intervention.
4. Patients with previous malignancies other than the target malignancy to be investigated in this trial
5. Known history of positive testing for Human Immunodeficiency Virus (HIV) or known Acquired Immune Deficiency Syndrome (AIDS)
6. Clinical or laboratory history or evidence of Hepatitis C Virus (HCV) or Hepatitis B Virus (HBV) indicating acute or chronic infection
7. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (> 10 mIU/mL)
8. Treatment with another investigational agent since the beginning of the screening period
9. Uncontrolled intercurrent illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2031-12-30 (Estimated)

PRIMARY OUTCOMES:
Phase I: Safety and tolerability (Adverse Event reported per CTCAE v5) | Up to 2 Years.
  Incidence of Adverse Event reported per CTCAE v5.
Phase I/II: Disease-Free Survival | Up to 2 years.
  Time from randomization to documented recurrence of disease.

SECONDARY OUTCOMES:
Phase I: Disease-Free Survival | Up to 2 Years.
  Time from randomization to documented recurrence of disease.
Phase I: Tumor response rate | Up to 2 years.
  Percentage of patients whose best overall response is either a Complete Response or a Partial Response according to RECIST version 1.1 criteria.
Phase I/II: Safety and tolerability (Adverse Event reported per CTCAE v5) | Up to 2 years.
  Incidence of Adverse Event reported per CTCAE v5.
Phase I/II: Distant Metastases-Free Survival | Up to 2 years.
  Time from randomization to documented first occurrence of distant metastasis.
Phase I/II: Loco-Regional Relapse-Free Survival | Up to 2 years.
  Time from randomization to documented loco-regional recurrence.
Phase I/II: Overall Response Rate in patients with recurrent disease | Up to 2 years.
  Percentage of patients with a best overall response of complete response or partial response according to RECIST, version 1.1 criteria.

CONTACTS AND LOCATIONS:
Locations (14):
- Mayo Clinic Jacksonville, Jacksonville, Florida, United States
- France (5):
  - Hôpital Saint André - CHU de Bordeaux, Bordeaux
  - Hôpital de la Timone, Marseille
  - Institut Curie, Paris
  - IUCT Toulouse, Toulouse
  - Institut Gustave Roussy, Villejuif
- Spain (6):
  - Hospital Universitari Vall d Hebrón, Barcelona
  - Institut Català d Oncologia - Hospital Duran i Reynals, Barcelona
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Málaga - Hospital Civil, Málaga
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela
- United Kingdom (2):
  - NHS Clatterbridge Cancer Center, Liverpool
  - Aintree University Hospital NHS Fondation Trust, Liverpool

IPD SHARING:
Plan to Share IPD: No